CLINICAL TRIAL: NCT05814367
Title: Clinical Investigation of Visual Acuity in Contact Lens Wearers After Instillation of Investigational Lubricating Eye Drops
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6503
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomized into the Test/Control sequence, to receive 1-2 drops on each eye (right eye followed by left eye) over soft spherical contact lenses, over two wear periods (test then control). A washout period of 90 minutes between eyedrop instillations will occur. The second eyedrop as per the randomization schedule will follow the same procedure as previously stated.
  Interventions: Drug: Blink® Tears eye drops in a multidose bottle; Drug: Preservative-free investigational lubricating eye drops in a Novelia® eyedropper
- Control/Test (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomized into the Control/Test sequence, to receive 1-2 drops on each eye (right eye followed by left eye) over soft spherical contact lenses, over two wear periods (control then test). A washout period of 90 minutes between eyedrop instillations will occur. The second eyedrop as per the randomization schedule will follow the same procedure as previously stated.
  Interventions: Drug: Blink® Tears eye drops in a multidose bottle; Drug: Preservative-free investigational lubricating eye drops in a Novelia® eyedropper

INTERVENTIONS:
Drug: Blink® Tears eye drops in a multidose bottle — Control
Drug: Preservative-free investigational lubricating eye drops in a Novelia® eyedropper — Test

SUMMARY:
This will be a single-visit, multi-site, randomized, single-masked, bilateral, active-controlled, non-dispensing, 2X2 crossover study.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

The subject must:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 69 (inclusive) years of age at the time of screening.
4. By self-report, habitually wear soft spherical contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e., not extended wear modality). Habitual wear is defined as a minimum of 6 hours per day, for a minimum of 2 days per week during the last 30 days.
5. Subjects must achieve visual acuity of 20/30 or better in each eye, with their habitual contact lenses.

Exclusion Criteria:

* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

The subject must not:

1. Be currently pregnant or lactating.
2. Be diabetic.
3. Be currently using any ocular medications or have any ocular infection of any type which may interfere with the clinical trial (at the investigator's discretion).
4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with the clinical trial, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g., rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g., SynergEyes, SoftPerm) within the past 3 months.
6. Have participated in any pharmaceutical or medical device related clinical trial within 14 days prior to study enrollment.
7. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
8. Be a current habitual user of prescription medication to treat dry eye and ocular discomfort, ocular steroids, or any medication (RX or OTC) except artificial tears, that would interfere with the clinical study (at the discretion of the investigator).
9. Have any known allergy or sensitivity to ingredients that the investigational product may contain (e.g., Sodium Chlorite, Boric Acid, Sodium Borate Decahydrate, Sodium Chloride, Potassium Chloride, Calcium Chloride Dihydrate, Magnesium Chloride Hexahydrate, Polyethylene Glycol 400, Sodium Hyaluronate and Purified Water).
10. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities, or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate participation or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
11. Have a history of strabismus or amblyopia.
12. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, cataract removal, retinal laser photocoagulation, etc.).
13. Have any significant corneal distortion due to previous contact lens wear, surgery, or pathology (At the discretion of the investigator).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (3):
- United States (3):
  - VRC, Jacksonville, Florida
  - Maitland Vision Center - North Orlando Ave, Maitland, Florida
  - Tyler Eye Associates, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 46 subjects were enrolled in this study. Of those enrolled, 44 subjects were dispensed at least one study lens, while 2 subjects failed to meet all eligibility criteria. All 44 dispensed subjects completed the study. 1-2 drops of Test and Control eye drops were administered to both eyes for every subject. This is a single visit study with 90-minute washout between period 1 and 2.
Groups:
- Test\Control: Subjects randomized to receive the Test Eye Drop in both eyes during the first period and the Control Eye Drop in both eyes during the second period
- Control\Test: Subjects randomized to receive the Control Eye Drop in both eyes during the first period and the Test Eye Drop in both eyes during the second period
Period: Period 1
Arm/Group | Test\Control | Control\Test
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test\Control | Control\Test
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dispensed Subjects: All subjects dispensed at least one study lens
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 5
  Black or African American | 8
  Native Hawaiian or Other Pacific Islander | 1
  White | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Monocular logMAR Visual Acuity
Description: Monocular visual acuity was measured at distance (4meter) using a logMAR (Logarithm of Minimal Angle of Resolution) scale under high luminance high contrast lighting conditions. VA was assessed using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. Letter-by-letter results calculated the visual acuity score for each chart read. LogMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 10 Minutes Post Eye Drop Administration
Population: All subjects who successfully complete all visits and do not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- Test: Subjects that received Test (Investigational) eye drop during either period of the study.
- Control: Subjects that received the Control eye drop during either period of the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 44 | 44
Number analyzed (Eyes) | 88 | 88
logMAR | 0.033 (0.1131) | 0.038 (0.1206)
Statistical Analysis 1: Comparison: Test vs Control; The sample size of 38 was calculated to provide at least 90% statistical power to test Non-inferiority of the Test lens compared to the Control lens using a paired t-test with a two-sided type I error rate of 5%; Test type: Non-Inferiority — A non-inferiority margin of 0.05 logMAR was used; Linear Mixed Model; Kenward and Roger Method was used for the denominator degrees of freedom; Least-square Mean Difference = -0.005, 95% CI 2-sided [-0.025 to 0.014], Standard Error of Mean 0.010 — Mean difference was calculated as Test minus Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; 1 day per subject
Description: All subjects dispensed a study lens.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT05814367/Prot_SAP_000.pdf